CLINICAL TRIAL: NCT06905600
Title: Transient Pseudohypoaldosteronism Affecting Children With Urinary Tract Malformation: Diagnosis and Management in a French Retrospective Study
Brief Title: Transient Pseudohypoaldosteronism Affecting Children With Urinary Tract Malformation
Acronym: TPHA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9139
Record Dates: First submitted 2024-07-08; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-07

CONDITIONS: Pseudohypoaldosteronism
Keywords: Pseudohypoaldosteronism; pseudohypoaldosteronism in children
MeSH Terms: conditions — Pseudohypoaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pseudohypoaldosteronism is a pathology affecting children under 6 months of age, little known but which can have serious consequences.

There are no real figures on the prevalence of this pathology in France. The exact pathophysiology is not known and the management is not currently codified.

This is why it is interesting to study this pathology and its treatment on a national scale in order to think about the best possible treatment, as well as to raise awareness of this pathology among different health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Minor subjects aged less than 6 years at the time of diagnosis
* Diagnosis of pseudohypoaldosteronism in the context of urinary malformation and/or urinary infection between January 1, 2018 and December 31, 2023
* Subject (and/or their parental authority) having not expressed, after information, their opposition to the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Subject (or their parents) having expressed their (their) opposition to participating in the study

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subjects aged less than 6 years at the time of diagnosis of pseudohypoaldosteronism in the context of urinary malformation and/or urinary infection between January 1, 2018 and December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
National comparison of clinical and therapeutic practices concerning the management of pseudohypoaldosteronism in children with urinary malformations and/or urinary infections | Up to 1 year
  This study compares clinical and therapeutic practices
  The retrospective analysis of the data will be carried out using classic statistical tests (Student's test, Fisher's test, ROC curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Service pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France